CLINICAL TRIAL: NCT01370876
Title: A Phase II Trial Evaluating Efficacy and Safety of Opatin® (Oxaliplatin)/5-FU in Patients With Recurrent or Metastatic Head and Neck Cancer
Brief Title: Efficacy and Safety Study of Oxaliplatin/5-FU in Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: company policy
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Cancer Center, Head and Neck Cancer Team, Taipei Mackay Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10CT006A
Record Dates: First submitted 2011-03-28; First posted 2011-06-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Cancer of the Head and Neck; Neoplasms, Head and Neck
Keywords: Oxaliplatin; Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin/5-FU (Experimental)
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin will be administered as a 2-hour infusion first on Day 1, followed by 5-FU i.v. infusion for 48 hours (Day 1 and Day 2), repeated every 2 weeks, 4 weeks as a cycle.
  Other Names: Opatin

SUMMARY:
To evaluate the objective response rate of oxaliplatin combined with 5-FU in patients with recurrent or metastatic head and neck cancer and to assess the safety profile of these treatment regimen.

DETAILED DESCRIPTION:
To evaluate the objective response rate of oxaliplatin combined with 5-FU in patients with recurrent or metastatic head and neck cancer.

To assess the safety profile of these treatment regimen. To evaluate the duration of response of oxaliplatin/5-FU.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been histologically confirmed squamous cell carcinoma of the head and neck (SCCHN) except nasopharyngeal cancer.
* Patients must have recurrent or metastatic disease and for which curative surgery or radiotherapy do not exist or are no longer effective.
* Prior to entering the protocol treatment, it has to be more than 6 months interval between previous systemic chemotherapy and protocol treatment.
* The disease must have been measurable by computed tomographic (CT) scan or MRI (done within 30 days of study entry) and the diameter of the target tumor is at least more than 1 cm.
* Patients must be 20 years of age and 75 years of age.
* Patients must have an ECOG performance status score 2.
* Patient's hematologic function, liver function and renal function must meet the eligibility requirements.
* Patients must sign the informed consent.

Exclusion Criteria:

* Patients with known hypersensitivity history to Platinum compounds or to 5-Fluorouracil.
* Patients with brain metastases.
* Patients with bone metastases only.
* Patients with pregnancy or breast-feeding.
* Patient with CTC (NCI Common Toxicity Criteria) grade 2 peripheral neuropathy of any cause that is clinically detectable.
* Patients who have serious concomitant illness that might be aggravated by chemotherapy and other conditions which will be judged by physician's discretion.
* Patients who are receiving other anticancer cancer drug(s) for SCCHN.

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate | every 12 weeks
  To evaluate the objective response rate of oxaliplatin combined with 5-FU in patients with recurrent or metastatic head and neck cancer

SECONDARY OUTCOMES:
Safety | Each patient will be followed for 30 days after the last dose of study medication
  To assess number of participants with adverse events of these treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Chang Yi Fan, M.D., Principal Investigator — Taipei Mackay Memorial Hospital
Locations (1):
- Taipei Mackay Memorial Hospital, Taipei, Taiwan